CLINICAL TRIAL: NCT06899074
Title: Evaluating the Effects of Omega-3 Polyunsaturated Fatty Acids in Pediatric Migraine Patients
Brief Title: Omega-3 Supplementation for Pediatric Migraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Nutrition Obesity Research Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 24-2715; P30DK056350 (NIH)
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Coconut Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple masking to allocation sequence. All subjects, the research personnel and the biostatistician will be masked to the allocation sequence. Only the dispensing pharmacist and the unmasked data manager are not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega 3 Polyunsaturated Fats (Experimental): Two in-person study visits (baseline, week 12) for collection of a blood sample, completion of validated questionnaires, and two 24-hour dietary recalls conducted over the phone
  Two study phone calls (week 4, week 8) to determine study adherence. Two additional study phone calls will be conducted to conduct 24-hour dietary recalls at baseline and week 12. All subjects (with the help of their parents) will complete a demographics form and headache/medication history form as part of the study's baseline procedures.
  A blood sample will be collected from all subjects at baseline and week 12 to determine whether the intervention increases omega-3 index in the blood via finger prick.
  Self-reported measures will be collected via survey.
  Post-baseline changes in migraine disability, psychological distress, and health-related quality of life will be assessed using validated self-reported questionnaires to compare the effects of omega-3 PUFA intervention versus placebo.
  Interventions: Dietary Supplement: Omega 3 Polyunsaturated Fats
- Matching Placebo (Placebo Comparator): Two in-person study visits (baseline, week 12) for collection of a blood sample, completion of validated questionnaires, and two 24-hour dietary recalls conducted over the phone
  Two study phone calls (week 4, week 8) to determine study adherence. Two additional study phone calls will be conducted to conduct 24-hour dietary recalls at baseline and week 12. All subjects (with the help of their parents) will complete a demographics form and headache/medication history form as part of the study's baseline procedures.
  A blood sample will be collected from all subjects at baseline and week 12 to determine whether the intervention increases omega-3 index in the blood via finger prick.
  Self-reported measures will be collected via survey.
  Post-baseline changes in migraine disability, psychological distress, and health-related quality of life will be assessed using validated self-reported questionnaires to compare the effects of omega-3 PUFA intervention versus placebo.
  Interventions: Other: Matching Placebo

INTERVENTIONS:
Dietary Supplement: Omega 3 Polyunsaturated Fats — Omega-3 PUFA dietary supplement daily for 12 weeks. The intervention is 1 teaspoon of liquid omega-3 containing oil profile 40% EPA / 60% DHA.
  Arms: Omega 3 Polyunsaturated Fats
Other: Matching Placebo — The placebo is a matched 1 teaspoon liquid of coconut oil, consisting mainly of saturated fatty acids and lacking omega-3 fatty acids.
  Other Names: Coconut oil
  Arms: Matching Placebo

SUMMARY:
The purpose of the study is to assess the biochemical and clinical effects of omega-3 polyunsaturated fatty acid (PUFA) supplementation in youth suffering from migraine, including its effects on migraine disability, psychological distress, and overall quality of life. This study duration 12 weeks.

DETAILED DESCRIPTION:
Omega-3 polyunsaturated fatty acids (PUFAs), particularly eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), hold potential therapeutic benefit for pediatric migraine due to their potent anti-inflammatory, anti-nociceptive, and neuromodulatory properties, which impact the pathophysiology of migraine. Dietary alteration and supplementation of omega-3 PUFAs have been shown to decrease the frequency, duration, and severity of headaches in adults with migraine, yet no rigorous clinical studies on omega-3 PUFA supplementation have been conducted in children and/or adolescents suffering from migraine. This study will establish feasibility of the intervention of omega-3 PUFA supplementation for pediatric migraine (i.e., provide proof-of-concept that the intervention raises omega-3 index levels compared to placebo).

The investigators will enroll 80 children and adolescents (ages 10-17 years) with a diagnosis of migraine and randomize participants 1:1 to receive an omega-3 PUFA dietary supplement intervention or placebo daily for 12 weeks, with assessments conducts at baseline and at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 10 and 17 years
* Parent consent and subject assent
* Diagnosis of migraine based on the third edition of the International Classification of Headache Disorders (ICHD-3) criteria

Exclusion Criteria:

* Known allergy to fish or seafood
* Current use of an omega-3 dietary supplement
* Significant neurological or psychiatric disorders or developmental delays
* Non-English speaking
* Allergy to coconut
* Pregnancy

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Omega-3 index levels in blood | Baseline and 12 weeks
  Compare the change in omega-3 index levels between the intervention and control groups via finger prick blood test.
Rate of self-reported pain intensity levels | Baseline and 12 weeks
  The associations between omega-3 index levels and pain intensity will be assessed based on validated self-report measures using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Pain Intensity Measure. The PROMIS Pain Intensity instruments assess how much the child hurts. The PROMIS Pediatric Pain Intensity Measure is a 3-item, self-report measure for children and adolescents ages 8 to 18 with chronic pain, using a 5-point Likert scale including three items rating pain from "Had no pain" = 1 to "Very severe" = 5. To find the total raw score for the short form, sum the values of the response to each question. For example, the lowest possible raw score is 3; the highest possible raw score is 15. All questions must be answered in order to produce a valid score. A lower score will indicate lower levels of pain intensity in the pediatric patient.
Rate of self-reported pain interference levels | Baseline and 12 weeks
  The associations between omega-3 index levels and pain interference will be assessed based on validated self-report measures using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Pain Interference Scale. The PROMIS Pediatric Pain Interference Scale is an 8-item self-report questionnaire completed by children that assesses how pain impacts a child's daily activities of living and the enjoyment of those activities using a 5-point likert scale. The PROMIS Pediatric Pain Interference Measure is a 3-item, self-report measure for children and adolescents ages 8 to 18 with chronic pain, using a 5-point Likert scale. This survey is measured on a scale of 0-4, from 0 being never to 4 being almost always. A lower score will indicate less pain interference in the pediatric patient.
Assess the effect of omega-3 PUFA intervention vs. placebo on migraine disability. | Baseline and 12 weeks
  The validated Pediatric Migraine Disability Assessment tool (PedMIDAS) will be used to measure migraine disability by self-report. PedMIDAS was developed to assess migraine disability in pediatric and adolescent patients ages 4-18. It is intended to be self-administered by the patient and their parent. The PedMIDAS is scored by summing the answers across 6 questions. If a range is provided as an answer, either use the high end of the range or prompt for a single answer. The grading scale for the PedMIDAS:
  PedMIDAS Score Range Disability Grade 0 to 10 Little to none 11 to 30 Mild 31 to 50 Moderate Greater than 50 Severe
Assess the effect of omega-3 PUFA intervention vs. placebo on psychological distress. | Baseline and 12 weeks
  The validated Revised Children's Anxiety and Depression Scale (RCADS)-short version 24 will be used to measure psychological distress by self-report. The RCADS is a 24-item self-report questionnaire designed to assess symptoms of anxiety and depression in children and adolescents aged 8 to 18 years using a 4-point Likert scale. Each item is assigned a numerical value from 0-3, where 0 = Never, 1 = Sometimes, 2 = Often, and 3 = Always, where a higher score indicates a higher level of anxiety and/or depression in the pediatric patient.
Assess the effect of omega-3 PUFA intervention vs. placebo on quality of life. | Baseline and 12 weeks
  The validated Pediatric Quality of Life Inventory 25 (PedsQL Inventory25) will be used to measure quality of life by self-report. The PedsQL Measurement Model is a modular approach to measuring health-related quality of life (HRQOL) assessed on a 4-point Likert scale. This survey is measured on a scale of 0-4, from 0 being never to 4 being almost always. The items in the PedsQL are designed to be reverse-scored (i.e. 0=100, 1=25. 2=50, 3=75, 4=0), meaning that higher scores on each item indicate a better experience or perception of certain area of health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Sawicki, DDS, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning at 12 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.